CLINICAL TRIAL: NCT03166644
Title: Individualized Goal-directed Sufentanil Administration Versus Standard Therapy in Patients Undergoing Major Abdominal Surgery: A Randomized Controlled Feasibility Trial.
Brief Title: Individualized Goal-directed Sufentanil Administration Versus Standard Therapy in Patients Undergoing Major Abdominal Surgery
Acronym: PHOENIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Rennes University Hospital (Other); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-335; 2016-001603-23 (Other: 2016-001603-23)
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2019-08

CONDITIONS: Major Abdominal Surgery
Keywords: Analgesia Nociception Index (ANI); Postoperative Analgesia; Postoperative Hypoxemia

STUDY DESIGN:
Intervention Model Description: Participants receive an intervention throughout the protocol
Who Masked: Participant
Masking Description: Simple Blind : participants are unaware of the intervention assignment; investigators are aware.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Patients with major abdominal surgery
  Interventions: Device: Analgesia Nociception Index (ANI)-guided sufentanil administration
- Intervention Group (Experimental): Patients with standard practice
  Interventions: Device: Analgesia Nociception Index (ANI)-guided sufentanil administration

INTERVENTIONS:
Device: Analgesia Nociception Index (ANI)-guided sufentanil administration — One recent observational study showed that ANI-guided remifentanil administration during vascular surgery resulted in low opioid consumption and low postoperative pain rates.

SUMMARY:
To determine whether a treatment strategy targeting an individualized sufentanil administration based on the Analgesia Nociception Index (ANI) could reduce the total dose of sufentanil during major abdominal surgery, as compared with standard practice.

DETAILED DESCRIPTION:
Postoperative respiratory complications are the second most frequent complications after surgery, and a major burden in health care. Postoperative hypoxemia, which is one of the most meaningful factors associated with poor patient outcomes, is common after general anesthesia with rates as high as 30-50% in patients after abdominal surgery, even among those undergoing uneventful procedures.

Risk factors for early postoperative hypoxemia, whether modifiable or not, are mainly related to the patient condition, the surgical procedure and the intraoperative anesthesia management strategy, especially the detrimental effects resulting from potential residual effects of anesthetic agents. There is, to date, only limited data on the incidence of postoperative hypoxemia resulting from excessive intraoperative opioid administration.

The Analgesia Nociception Index (ANI) is a unit-less index ranging from 0 to 100 calculated from the instantaneous wavelet transform analysis of heart rate variability, which indirectly reflects the parasympathetic tone, with higher ANI values indicating a prominent parasympathetic tone. ANI is sensitive to nociception stimuli and has recently been proposed to evaluate the analgesia/nociception equilibrium. The few interventional studies that have investigated the ability of a protocol-driven intraoperative analgesia procedure to reduce postoperative pain have used mixed results. One recent observational study showed that ANI-guided remifentanil administration during vascular surgery resulted in low opioid consumption and low postoperative pain rates. In addition, to our knowledge, no study has investigated whether ANI monitoring can be used to improve postoperative outcome. Accordingly, to determine the impact of an ANI-guided individualized opioids administration on postoperative outcomes, a large multicenter randomized controlled trial is needed. However, before such a trial can take place, it is necessary to determine the feasibility in potential participating sites of successfully reducing intraoperative opioid consumption while reducing postoperative pain.

The purpose of this study was to examine the feasibility of undertaking such a trial. Our primary hypothesis is that individualizing sufentanil administration to target ANI values between 50 and 70 during major abdominal surgery could reduce the intraoperative dose of sufentanil, as compared with standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective major abdominal surgery
* Estimated duration of surgery greater than 2 hours

Exclusion Criteria:

* Emergency abdominal surgery
* Atrial fibrillation
* Patient with pacemaker
* Patient with heart transplant
* Chronic beta-blockade
* Intrathecal anesthesia
* Conditions affecting SpO2 measurement (e.g., methemoglobinemia)
* Morbid obesity (BMI> 35 kg/m2)
* Obstructive sleep apnea (OSA)
* Person under legal guardianship or curatorship
* No affiliation with the French health care system
* Pregnant or breastfeeding women
* Refusal to participate or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Total dose of sufentanil administered during major abdominal surgery | at day 0

SECONDARY OUTCOMES:
Percentage of time spent in the therapeutic target | at day 0
  (ANI between 50 and 70 for an energy between 0.05 and 2.5)
Number of patients with early postoperative hypoxemia | at 30 min, 1 hour, 2 hour and 3 hour after tracheal extubation
  (defined as SpO2 <94% in ambient air but responding to administration of oxygen by nasal cannula or facial mask)
Number of patients with late postoperative hypoxemia | at day 1 and 2 after surgery
  (defined as SpO2 <94% in ambient air but responding to administration of oxygen by nasal cannula or facial mask)
Time to extubation | at day 0
Need for postoperative oxygen therapy | at day 0
Postoperative pain score | at 30 min, 1 hour, 2 hour and 3 hour after extubation
  evaluated by a visual numeric scale (EVN) at rest and after exercise
Postoperative pain score | on postoperative Day 1 and Day 2
  evaluated by a visual numeric scale (EVN) at rest and after exercise
Total dose of morphine administered in postoperative care unit | at day 1
  PACU
Duration of PACU stay | at day 1
  defined by the time interval to reach an Aldrete score of 9 or more after the end of sufentanil administration

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel FUTIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France